CLINICAL TRIAL: NCT06726304
Title: A Pilot Intervention Study to Increase Physical Contact Between Prenatally Anxious/Depressed Mothers and Their Infants to Improve Maternal Sensitivity
Brief Title: Increasing Physical Contact Between Prenatally Anxious/Depressed Mothers and Their Infants to Improve Maternal Sensitivity.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Brain Canada (Other)
Responsible Party: Principal Investigator, Eszter Szekely, Co-Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024-989
Record Dates: First submitted 2024-12-01; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Prenatal Anxiety; Prenatal Depression; Maternal Sensitivity
Keywords: baby carrier; maternal sensitivity; inter-personal neural synchrony; perinatal anxiety; perinatal depression

STUDY DESIGN:
Intervention Model Description: Behavioural intervention with rolling recruitment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baby Carrier Intervention Group (Experimental): Participants and their babies will be visited twice by trained research staff in their home. Once at the beginning of the study (at 8 weeks postpartum) and for a second time at the end of the study (at 16 weeks postpartum). During the first visit, mothers will choose between two soft ergonomic baby carriers and be given instructions regarding the expected frequency and length of usage. Maternal sensitivity will be observed during a 15-minute free play session of the mother-baby dyad. During the second home visit, inter-personal neural synchrony in mother-baby dyads will be assessed during a joint attention task (9 minutes). Participants will also be interviewed about their lived experiences with babywearing and increased physical contact with their baby (30-40 minutes). Finally, participants will complete questionnaires about mother-infant bonding, depression and anxiety symptoms, and rate the burden of the protocol.
  Interventions: Behavioral: Baby Carrier Intervention
- Waitlist Control Group (No Intervention): The waitlist control group will be assessed using the same measures as the intervention group (described above) except for the open-ended interview questions about their lived experiences with regular babywearing and increased physical contact with their baby.
  At the end of the second home visit, all waitlist control participants will be offered to choose between the same two ergonomic baby carrier models as the intervention group, and will be provided with the same instructions regarding the recommended frequency and length of use as intervention group participants at the beginning of the study.

INTERVENTIONS:
Behavioral: Baby Carrier Intervention — Mothers in the intervention group will have the opportunity to choose between two different soft ergonomic baby carriers and will receive instructions on how to use the carrier of their choice. Infants will be placed chest-to-chest in the carrier, supported by the mother's upper torso for a prescribed amount of time during the period of six weeks.
  Arms: Baby Carrier Intervention Group

SUMMARY:
The goal of this randomized controlled pilot trial is to evaluate the feasibility, acceptability, and clinical utility of a baby carrier intervention aimed at improving maternal sensitivity and mother-infant bonding in prenatally anxious/depressed mothers. The study has three main questions:

1. Is the intervention feasible (e.g., enrollment and recruitment rates) and acceptable to participants (e.g., compliance and perceived benefits)?
2. Does the intervention improve maternal sensitivity compared to a waitlist control group?
3. Does the intervention increase mother-infant neural synchrony compared to a waitlist control group, measured using functional near-infrared spectroscopy?

Participants will A. Choose between two soft ergonomic baby carriers and be expected to use the baby carrier for the prescribed amount of time (intervention group).

B. Have two home visits, one at the start (at postpartum week 8) and another one at the end of the study (at postpartum week 16).

C. Complete questionnaires about depression and anxiety symptoms, mother-infant bonding, and rate protocol burden.

D. Share their feelings and lived experiences about the frequent use of a baby carrier and increased physical contact with their baby through open-ended interview questions (intervention group).

DETAILED DESCRIPTION:
The intervention involves mothers in the experimental group using a soft ergonomic baby carrier for a prescribed amount of time over a period of six weeks. Weekly adherence self-reports will be collected via REDCap. Participants will be recruited from the Perinatal Multisite Databank (PMD), an ongoing clinical cohort of individuals receiving psychiatric services during pregnancy and the first six months postpartum in the province of Quebec, Canada.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* be able to communicate in English or French
* diagnosed with a depressive or anxiety disorder (or both) during their intake visit within the Perinatal Multisite Databank (PMD)
* residing in the greater Montreal area
* have given birth to a healthy baby

Exclusion Criteria:

* having known alcohol or substance use issues,
* having been diagnosed with psychosis or schizophrenia during the PMD intake assessment, or have had thoughts of harming the self or the baby
* having physical restrictions that may prevent the regular use of a baby carrier
* taking any medications regularly that cause potential participants to feel drowsy or dizzy
* already using a baby carrier with their current baby for more than 5 hours a week

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Proportion of Eligible Participants Successfully Enrolled and Retained Over 12 Months | From the beginning of recruitment to the end of the last assessment (at 16 weeks postpartum)
  To assess the feasibility of the baby carrier intervention, including recruitment, enrollment, and retention rates, using the ratio of eligible versus enrolled participants and enrolled versus retained participants.

SECONDARY OUTCOMES:
Acceptability: Adherence to the baby carrier intervention | From the beginning of the intervention (at 8 weeks postpartum) to the end of the intervention (up until 16 weeks postpartum)
  Acceptability will be evaluated based on i) compliance with the prescribed length of baby carrier usage according to self-reports, ii) rating the burden of the protocol low-moderate, and iii) report benefits associated with babywearing in the interview.

OTHER OUTCOMES:
Utility of the baby carrier intervention | From baseline assessment (at week 8) to final assessment (at week 16) of maternal sensitivity
  Utility of the baby carrier intervention will be evaluated by comparing the increase in maternal sensitivity scores from pre- to post-intervention between the intervention and control groups. Maternal sensitivity will be observed and rated using the Ainsworth's Maternal Sensitivity scales-a gold standard in the assessment of sensitive parenting- during a 15-minute free play session (5-minute without toys, 10-minute with toys). The play session will be recorded. Recordings will be coded by blinded and trained observers.
Inter-personal Neural Synchrony | During the second home visit (at week 16 postpartum)
  Inter-personal neural synchrony between mother and baby will be measured during the second home visit using non-invasive functional near-infrared spectroscopy (fNIRS), while the mother and baby complete a 6-minute still-face paradigm and a 3-minute joint video attention task. Prefrontal cortical activity will be captured across four regions (frontal/medial left/right) and compared between the intervention and control groups.
Qualitative Analysis of Maternal Experiences with Babywearing | During the second home visit (at week 16 postpartum)
  During the second home visit, open-ended interviews will be conducted with intervention group participants to explore their feelings and lived experiences about regular use of a baby carrier and increased physical contact with their baby. Sample questions cover usage frequency, circumstances, feelings, and likes/dislikes about babywearing. Interviews will be recorded unless participants opt out, transcribed verbatim, and analyzed using inductive content analysis. Transcription will be performed by a trained student under a signed non-disclosure agreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Davis Institute of the Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No